CLINICAL TRIAL: NCT05528276
Title: Does Preputial Inlay Graft Improves the Outcome of Tubularized Incised Plate Repair for Primary Distal Hypospadias? a Prospective Randomized Controlled Trial.
Brief Title: Does Graft Improves the Outcome TIP Repair for Primary Distal Hypospadias?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrahman Mohamed Abdelkader, teaching assistant of urology & andrology, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: hypospadias repair
Record Dates: First submitted 2022-08-28; First posted 2022-09-06 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Penile Hypospadias
MeSH Terms: conditions — Hypospadias | interventions — Sutureless Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard Tubularized incised plate urethroplasty (sTIPU) (Active Comparator)
  Interventions: Procedure: Repair surgery
- Preputial inlay graft urethroplasty (PIGU) (Active Comparator)
  Interventions: Procedure: Repair surgery

INTERVENTIONS:
Procedure: Repair surgery — 1. a circumscribing skin incision was made 2 mm below the hypospadias meatus,
  2. penile degloving,
  3. the para-urethral plate incision was made,
  4. A vertical midline incision of the urethral plate was made from within the hypospadiac meatus and extended up to the mid-glans.
  5. The urethral plate was tubularised, beginning proximally, and closed in two layers using 6/0 polyglactin 910 suture.
  6. The neomeatus was formed on a catheter 2 F larger than the urethral stent.
  7. A flap was harvested from the prepuce to cover the neourethra and finally glanuloplasty.
  8. A suitable urethral stent was left in situ for 7-10 days, with a compressive dressing applied.
     * Grafted tubularised incised-plate .
  1.Same steps but adding a graft (dorsal inlay) , 2. The graft will be taken from the inner preputial skin . 3. The graft will be sutured to overlying plate incision line from the old meatus to the tip of the glans.

SUMMARY:
Hypospadias is a common congenital anomalies in male children affecting 1 in 200-300 male births, the penis urethral opening is found ventrally, penile curvature and a lack of foreskin (1). Multiple operations are described , Tubularised incised-plate is the preferred option for distal hypospadias and with trial to extend the operation indication to proximal and redo hypospadias (2). Its simple operative technique made TIP repair gain worldwide acceptance in addition to the low complication rate & good cosmetic outcome (3).It has several complication as stenosis meatus, fistula formation , uretheral stricture and failed repair (4). Objective scoring systems were introduced to allow better judgment and identification of the postoperative results, depending on pre-operative and intra-operative criteria (5). Modifications of the T.I.P operation was done to reduce complication and allow better results by using a graft , Snodgraft vs Snodgrass operation are nearly equal regarding the outcomes (6). To our knowledge there is no definite recommendation.

ELIGIBILITY:
Inclusion Criteria:

1. Children age more than 12 months to 12 years.
2. De-novo penile hypospadias after degloving of penis intraoperative (fresh, not previously operated)

Exclusion Criteria:

1. Circumcised
2. Ventral Penile curvature ≥30° after penile degloving & artificial erection, (requiring transection of urethral plate).
3. Uretheral plate less than 6mm
4. Megameatus intact prepuce
5. Albumin less than 3.5 g/dL

Ages: 1 Year to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 25 (Estimated)
Dates: Start 2022-08-29 (Estimated); Primary Completion 2024-10-29 (Estimated); Study Completion 2024-10-29 (Estimated)

PRIMARY OUTCOMES:
Operation time. | intraoperative
  the duration of the operation will be measured from the start of anesthesia to end.
blood loss. | one hour postoperatively
  the amount of blood loss will be measured by CBC
site of the meatus | 6 months from the operation
  the meatal position will be measured in centimeters from the original position .

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alshafei A, Cascio S, Boland F, O'Shea N, Hickey A, Quinn F. Comparing the outcomes of tubularized incised plate urethroplasty and dorsal inlay graft urethroplasty in children with hypospadias: a systematic review and meta-analysis. J Pediatr Urol. 2020 Apr;16(2):154-161. doi: 10.1016/j.jpurol.2020.01.009. Epub 2020 Jan 22. PMID 32061491
- [Background] Liu MM, Holland AJ, Cass DT. Assessment of postoperative outcomes of hypospadias repair with validated questionnaires. J Pediatr Surg. 2015 Dec;50(12):2071-4. doi: 10.1016/j.jpedsurg.2015.08.047. Epub 2015 Sep 1. PMID 26455467
- [Background] Pfistermuller KL, McArdle AJ, Cuckow PM. Meta-analysis of complication rates of the tubularized incised plate (TIP) repair. J Pediatr Urol. 2015 Apr;11(2):54-9. doi: 10.1016/j.jpurol.2014.12.006. Epub 2015 Feb 26. PMID 25819601
- [Background] Seleim HM, ElSheemy MS, Abdalazeem Y, Abdullateef KS, Arafa MA, Shouman AM, Elsaket H, Kaddah SN, Elbarbary MM. Comprehensive evaluation of grafting the preservable narrow plates with consideration of native plate width at primary hypospadias surgery. J Pediatr Urol. 2019 Aug;15(4):345.e1-345.e7. doi: 10.1016/j.jpurol.2019.05.002. Epub 2019 May 9. PMID 31155410
- [Background] Ahmed M, Alsaid A. Is combined inner preputial inlay graft with tubularized incised plate in hypospadias repair worth doing? J Pediatr Urol. 2015 Aug;11(4):229.e1-4. doi: 10.1016/j.jpurol.2015.05.015. Epub 2015 Jun 12. PMID 26119452